CLINICAL TRIAL: NCT02289404
Title: Clinical Trial to Evaluate the Food Effect on the Pharmacokinetics of NVP-1203 in Healthy Adult Subjects
Brief Title: A Study to Evaluate the Food Effect on the Pharmacokinetics of NVP-1203
Acronym: NVP-1203
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NVP Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NVP-1203_FE
Record Dates: First submitted 2014-11-09; First posted 2014-11-13 (Estimated); Last update posted 2019-03-08 (Actual); Status verified 2019-03

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NVP-1203(fed then fasting) (Experimental): Subjects will receive a oral dose of NVP-1203 under fed conditions in period 1, then subjects will receive a oral dose of NVP-1203 under fasting conditions in period 2
  Interventions: Drug: NVP-1203
- NVP-1203(fasting then fed) (Experimental): Subjects will receive a oral dose of NVP-1203 under fasting conditions in period 1, then subjects will receive a oral dose of NVP-1203 under fed conditions in period 2
  Interventions: Drug: NVP-1203

INTERVENTIONS:
Drug: NVP-1203 — Oral
  Arms: NVP-1203(fed then fasting)
Drug: NVP-1203 — Oral
  Arms: NVP-1203(fasting then fed)

SUMMARY:
The purpose of this study is to evaluate food effect on the pharmacokinetics of NVP-1203

DETAILED DESCRIPTION:
This study is designed as randomized, open-label, crossover assignment for evaluate the food effect on the pharmacokinetics of NVP-1203 in healthy adult subjects

ELIGIBILITY:
Inclusion Criteria:

* healthy adult subjects who signed informed consent

Exclusion Criteria:

* Subjects has a history of allergy reaction of study drug ingredient
* Subjects participated in another clinical trial within 3 months prior to administration of the study drug
* Inadequate subject for the clinical trial by the investigator's decision

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2019-01-18 (Actual); Primary Completion 2019-01-27 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics : Cmax | 0-24 hours
  Maximum plasma concentration
Pharmacokinetics : AUCt | 0-24 hours
  Area under the concentration-time curve

SECONDARY OUTCOMES:
Pharmacokinetics : AUCinf | 0-24 hours
  AUC extrapolated to infinity
Pharmacokinetics : Tmax | 0-24 hours
  Time to reach the Cmax
Pharmacokinetics : t1/2 | 0-24 hours
  Terminal elimination half-life

CONTACTS AND LOCATIONS:
Overall Officials: Yoon Y Ran, M.D., Principal Investigator — Kyungpook National University Hospital
Locations (1):
- Kyungpook National University Hospital, Daegu, Dongdeok-ro, South Korea

IPD SHARING:
Plan to Share IPD: No